CLINICAL TRIAL: NCT07315620
Title: Evaluation of Passive Fit in Implant-Supported Complete-Arch Prostheses Using Three Digital Workflows, Including an Automated AI-Assisted Protocol: A Randomized Clinical Trial
Brief Title: Passive Fit of Implant-Supported Complete-Arch Prostheses Using Digital Workflows
Acronym: MFS03-Pdental
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Miguel Gómez Polo, Associate Professor of Prosthodontics, Department of Conservative Dentistry and Prosthodontics, Faculty of Dentistry, Universidad Complutense de Madrid, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25/701-IC_P_CE
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Prosthesis and Implant Dentistry
Keywords: Implant-Supported Prosthesis; Full-Arch Rehabilitation; Passive Fit; Digital Workflow; Computer-Aided Design and Manufacturing (CAD/CAM); AI-Assisted Workflow

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group interventional clinical trial. Eligible participants are randomly assigned in a 1:1:1 ratio to one of three independent study arms, each corresponding to a different digital workflow for the fabrication of a definitive full-arch implant-supported prosthesis. Each participant receives a single definitive prosthesis fabricated using the assigned workflow, and outcomes are assessed once at the time of definitive prosthesis placement.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBCT-STL Alignment (Medicalfit 1.0) (Active Comparator): Participants in this arm will receive a definitive, screw-retained, implant-supported full-arch prosthesis fabricated using a digital workflow based on manual alignment of CBCT and intraoral scan (STL) datasets. Scannable healing abutments (Tissue Shapers-IF; MedicalFit, Úbeda, Spain) will be connected to multi-unit abutments according to the manufacturer's instructions. An intraoral scan and a CBCT scan will be obtained and manually aligned by the operator during the CAD design stage using reference points visible in both datasets. Prosthetic framework passivation is performed manually during the CAD phase. The definitive prosthesis is designed and manufactured using CAD/CAM technology in monolithic zirconia (IPS e.max ZirCAD Prime; Ivoclar, Schaan, Liechtenstein). This workflow is fully operator-dependent and serves as an active comparator.
  Interventions: Procedure: CBCT-STL Alignment Workflow
- Splint-Guided Alignment (Medicalfit 2.0) (Active Comparator): Participants in this arm will receive a definitive, screw-retained, implant-supported full-arch prosthesis fabricated using a digital workflow that incorporates a rigid reference splint with metallic abutment cylinders to assist manual dataset alignment. Scannable healing abutments (Tissue Shapers-IF; MedicalFit, Úbeda, Spain) are connected to multi-unit abutments. A calibrated rigid splint is intraorally adapted and connected to the abutment cylinders, and both intraoral and splint scans are obtained. The acquired datasets are imported into CAD software, where CBCT-STL registration is performed manually using the splint as a reference. The definitive prosthetic framework is designed and manufactured using CAD/CAM technology in monolithic zirconia (IPS e.max ZirCAD Prime; Ivoclar, Schaan, Liechtenstein). This workflow remains operator-dependent and serves as an active comparator.
  Interventions: Procedure: Splint-Guided Alignment Workflow
- Automated AI-Assisted CBCT-STL Alignment (Medicalfit 3.0) (Experimental): Participants in this arm will receive a definitive, screw-retained, implant-supported full-arch prosthesis fabricated using an automated AI-assisted digital workflow. Scannable healing abutments (Tissue Shapers-IF; MedicalFit, Úbeda, Spain) are connected to multi-unit abutments according to the manufacturer's protocol. An intraoral scan and a CBCT scan are acquired and imported into dedicated AI-assisted software (Pdental; MedicalFit, Úbeda, Spain). The software automatically detects the scan bodies and performs CBCT-STL dataset alignment prior to CAD/CAM prosthesis fabrication. The definitive prosthesis is designed and manufactured using CAD/CAM technology in monolithic zirconia (IPS e.max ZirCAD Prime; Ivoclar, Schaan, Liechtenstein). This workflow minimizes operator involvement and represents the experimental intervention.
  Interventions: Procedure: Automated AI-Assisted CBCT-STL Alignment Workflow

INTERVENTIONS:
Procedure: CBCT-STL Alignment Workflow — This procedure consists of a fully digital workflow for fabricating a screw-retained, implant-supported full-arch prosthesis using manual alignment between CBCT and intraoral scan (STL) data. Scannable healing abutments (Tissue Shapers-IF; MedicalFit, Úbeda, Spain) are attached to multi-unit abutments torqued to 10 Ncm. A CBCT scan and an intraoral scan are acquired and manually aligned in CAD software using operator-defined reference points. Passive fit is adjusted manually during the CAD design stage. The definitive framework is milled from monolithic zirconia (IPS e.max ZirCAD Prime; Ivoclar, Schaan, Liechtenstein). This workflow is operator-dependent and serves as the control procedure.
  Arms: CBCT-STL Alignment (Medicalfit 1.0)
Procedure: Splint-Guided Alignment Workflow — This procedure employs a rigid reference splint with metallic abutment cylinders to guide dataset alignment for full-arch prosthesis fabrication. Scannable healing abutments (Tissue Shapers-IF; MedicalFit, Úbeda, Spain) are connected to multi-unit abutments torqued to 10 Ncm. The splint is attached intraorally and scanned extraorally to capture implant positions. The splint and intraoral scans (STL) are imported into CAD software, where manual alignment is performed using the splint as a reference. The final monolithic zirconia framework (IPS e.max ZirCAD Prime; Ivoclar, Schaan, Liechtenstein) is designed and milled via CAD/CAM. This workflow is operator-dependent and used as an active comparator.
  Arms: Splint-Guided Alignment (Medicalfit 2.0)
Procedure: Automated AI-Assisted CBCT-STL Alignment Workflow — This procedure uses AI-assisted software (Pdental, MedicalFit, Úbeda, Spain) to automate the alignment of CBCT and intraoral scan (STL) datasets for full-arch prosthesis fabrication. After placement of scannable healing abutments (Tissue Shapers-IF; MedicalFit), intraoral and CBCT scans are obtained. The software automatically detects healing abutments, performs CBCT-STL registration, and corrects deviations greater than 120 µm to achieve passive fit within clinically acceptable limits. The corrected digital model is exported in STL format for CAD design and CAM milling of a monolithic zirconia screw-retained prosthesis (IPS e.max ZirCAD Prime; Ivoclar, Schaan, Liechtenstein). This workflow minimizes operator dependency based on an AI-assisted automation. .
  Arms: Automated AI-Assisted CBCT-STL Alignment (Medicalfit 3.0)

SUMMARY:
The goal of this clinical trial is to evaluate and compare three digital workflows for the fabrication of definitive implant-supported full-arch prostheses in adult patients requiring fixed implant rehabilitation.

The main questions it aims to answer are:

* Does an automated AI-assisted digital workflow improve the passive fit of definitive full-arch implant-supported prostheses compared with manual and splint-guided alignment workflows?
* Are there differences in marginal, geometric, mechanical, and radiographic passivity among the three digital workflows? Researchers will compare manual CBCT-STL alignment, splint-guided alignment, and automated AI-assisted CBCT-STL alignment to see if the degree of digital workflow automation affects the passive fit of definitive full-arch implant-supported prostheses.

Participants will:

* Be adults (18 years and older) indicated for fixed implant-supported full-arch rehabilitation.
* Receive a definitive, screw-retained, full-arch implant-supported prosthesis fabricated using one of the three assigned digital workflows.
* Undergo standardized clinical and radiographic assessments at the time of definitive prosthesis placement to evaluate prosthesis passive fit.

DETAILED DESCRIPTION:
This randomized controlled clinical trial aims to evaluate and compare the passive fit of definitive full-arch implant-supported prostheses fabricated using three different digital workflows with increasing levels of automation for implant position registration and prosthesis fabrication.

Full-arch implant-supported rehabilitations require a high level of precision to ensure passive fit between the prosthetic framework and the implant-abutment connections. Inadequate passive fit may lead to mechanical complications, biological overload, or long-term prosthetic failure. Digital workflows combining intraoral scanning (IOS) and cone-beam computed tomography (CBCT) have been introduced to improve accuracy; however, differences in data acquisition and dataset alignment strategies may influence the final prosthetic fit.

The study will include adult patients (18 years and older) indicated for fixed implant-supported full-arch rehabilitation in the maxilla or mandible. Eligible participants will be recruited from the Faculty of Dentistry of the Complutense University of Madrid and associated clinical centers. After providing written informed consent, participants will be randomly assigned in a 1:1:1 ratio to one of three digital workflows:

1. Manual CBCT-STL alignment (MedicalFit 1.0): implant positions are obtained by combining intraoral scans and CBCT data, with dataset registration performed manually by the operator based on visual alignment of scan bodies.
2. Splint-guided alignment (MedicalFit 2.0): a calibrated rigid reference splint with metallic cylinders is used to stabilize implant positions and assist manual dataset registration, aiming to reduce operator-dependent variability.
3. Automated AI-assisted CBCT-STL alignment (MedicalFit 3.0 - Pdental): dataset registration and passivation are performed automatically by dedicated software using advanced algorithms for implant detection and alignment, without manual intervention.

All participants will receive a definitive, screw-retained, full-arch implant-supported prosthesis fabricated according to the assigned digital workflow. Prosthetic materials and clinical procedures will follow standard clinical practice. No outcome measures will be assessed during provisional prosthetic phases.

Passive fit will be evaluated exclusively at the time of definitive prosthesis placement using a standardized multi-assessment clinical approach performed at each implant-prosthesis connection.

Marginal passive fit will be assessed clinically by direct inspection using a calibrated periodontal probe. The presence or absence of marginal discrepancies between the prosthesis and the transepithelial abutment will be evaluated based on visual and tactile criteria, including the ability of the probe to penetrate the prosthesis-abutment interface.

Geometric passive fit will be evaluated using the modified Sheffield test. With all prosthetic screws loosened except for one distal screw, the presence of any lifting or separation of the prosthetic framework at the non-tightened connections will be assessed visually and tactually using an explorer probe.

Mechanical passive fit will be assessed through the tactile sensitivity of the passive screw test. Resistance perceived during screw tightening will be evaluated qualitatively to identify the presence of internal stresses or framework flexure during seating of the definitive prosthesis.

Radiographic passive fit will be assessed by measuring marginal gaps at the prosthesis-abutment interface on standardized periapical radiographs. Radiographic gaps will be quantified and classified using predefined ordinal thresholds to identify clinically relevant discrepancies.

Each assessment will be scored using an ordinal scale (0-2) based on predefined clinical criteria. To reflect clinical decision-making and ensure a conservative interpretation of prosthetic fit, a hierarchical aggregation rule will be applied. For each assessment dimension, the prosthesis-level score will be defined as the worst score observed among all implant-prosthesis connections. The global multi-assessment passive fit score (0-2) will then be defined as the worst score observed across all assessment dimensions.

Accordingly, if any implant-prosthesis connection exhibits a clinically relevant misfit in any assessment, the definitive prosthesis will be classified as non-passive. This approach reflects the clinical principle that lack of passive fit at a single connection compromises the overall prosthetic outcome.

The primary objective of the study is to determine whether increased automation in digital workflows improves the passive fit of definitive full-arch implant-supported prostheses. Secondary objectives include comparing marginal, geometric, mechanical, and radiographic passivity outcomes among the three workflows and exploring the relationship between workflow automation and prosthetic adaptation accuracy.

The study follows CONSORT guidelines and aims to provide clinically relevant evidence to support the optimization of digital workflows in full-arch implant-supported prosthetic rehabilitation

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older.
2. Patients indicated for fixed implant-supported full-arch rehabilitation in the maxilla or mandible.
3. Presence of clinically stable, osteointegrated titanium implants suitable for prosthetic rehabilitation.
4. Absence of clinical or radiographic signs of peri-implant disease.
5. Ability to understand the study procedures and provide written informed consent.
6. Willingness and ability to attend all required clinical visits and evaluations.

Exclusion Criteria:

1. Presence of peri-implant mucositis or peri-implantitis at the time of evaluation.
2. Implant mobility or implant positioning that prevents proper prosthetic rehabilitation.
3. Uncontrolled systemic medical conditions that could interfere with study participation or prosthetic treatment.
4. Cognitive, psychological, or medical conditions that limit the ability to comply with study procedures.
5. Inability to complete the required clinical evaluations or follow the study protocol, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Multi-assessment global passive fit score of definitive full-arch implant-supported prostheses | At definitive prosthesis placement
  Passive fit of the definitive full-arch implant-supported prosthesis will be evaluated using a standardized multi-assessment clinical approach. Marginal, geometric (modified Sheffield test), mechanical (passive screw test sensitivity), and radiographic passive fit will be assessed independently at each implant-prosthesis connection.
  Each assessment will be scored using an ordinal scale (0-2) based on predefined clinical criteria:
  0 = no detectable discrepancy, indicating adequate passive fit;
  1 = minor discrepancy, indicating a cl To obtain the prosthesis-level outcome, a conservative aggregation rule will be applied: for each assessment dimension, the prosthesis score will be defined as the worst score observed among all implant-prosthesis connections. The global multi-assessment passive fit score (0-2) will then be defined as the worst score observed across all assessment dimensions.

SECONDARY OUTCOMES:
Clinical marginal passive fit (probe assessment) | At definitive prosthesis placement
  Marginal passive fit will be evaluated clinically by direct inspection using a calibrated probe to assess the presence of marginal discrepancies between the prosthesis and the transepithelial abutment. Outcomes will be recorded using an ordinal scale (0-2) based on visual and tactile criteria defined as follows:
  0 = no visible gap and no probe penetration;
  1. = visible marginal discrepancy without probe penetration;
  2. = clinically detectable gap with probe penetration or visually, indicating lack of passive fit.
Radiographic marginal gap at the prosthesis-abutment interface | At definitive prosthesis placement
  Marginal gaps between the definitive prosthesis and the transepithelial abutment will be evaluated on standardized periapical radiographs. Measured gaps will be classified using an ordinal scale (0-2) as follows:
  0 = gap < 100 µm;
  1. = gap between 100 and 130 µm;
  2. = gap > 130 µm, indicating a clinically relevant misfit.
Geometric passive fit assessed by the modified Sheffield test | At definitive prosthesis placement
  Geometric passive fit will be evaluated using the modified Sheffield test by tightening a single distal prosthetic screw and assessing the presence of lifting or separation at the non-tightened implant-prosthesis connections. Outcomes will be classified as follows:
  0 = no visible or tactile separation;
  1. = slight visible separation without probe penetration;
  2. = clear separation with probe penetration, indicating absence of passive fit.
Mechanical passive fit assessed by passive screw test sensitivity | At definitive prosthesis placement
  Mechanical passive fit will be evaluated qualitatively based on tactile resistance perceived during tightening of the prosthetic screws. Outcomes will be classified using an ordinal scale (0-2) defined as follows:
  0 = smooth screw tightening without perceptible resistance;
  1. = mild or transient resistance without need for force;
  2. = clear resistance or framework flexure during tightening, indicating internal stress and lack of passive fit.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Gómez Polo, DDS, PhD, Study Director — School of Dentistry, Complutense University of Madrid. Pza Ramon y Cajal S/N. 28040 Madrid, Spain
Locations (1):
- University Complutense of Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations. The data collected include detailed clinical and radiographic information that could potentially allow re-identification of participants, even after de-identification. Data will be used solely for the purposes defined in the approved study protocol.

REFERENCES:
- [Background] Abduo J, Judge RB. Implications of implant framework misfit: a systematic review of biomechanical sequelae. Int J Oral Maxillofac Implants. 2014 May-Jun;29(3):608-21. doi: 10.11607/jomi.3418. PMID 24818199
- [Background] Heckmann SM, Karl M, Wichmann MG, Winter W, Graef F, Taylor TD. Cement fixation and screw retention: parameters of passive fit. An in vitro study of three-unit implant-supported fixed partial dentures. Clin Oral Implants Res. 2004 Aug;15(4):466-73. doi: 10.1111/j.1600-0501.2004.01027.x. PMID 15248882
- [Background] Abdelrehim A, Etajuri EA, Sulaiman E, Sofian H, Salleh NM. Magnitude of misfit threshold in implant-supported restorations: A systematic review. J Prosthet Dent. 2024 Sep;132(3):528-535. doi: 10.1016/j.prosdent.2022.09.010. Epub 2022 Nov 7. PMID 36357194
- [Background] Pan Y, Tsoi JKH, Lam WYH, Pow EHN. Implant framework misfit: A systematic review on assessment methods and clinical complications. Clin Implant Dent Relat Res. 2021 Apr;23(2):244-258. doi: 10.1111/cid.12968. Epub 2020 Dec 16. PMID 33331058
- [Background] Gomez-Polo M, Alvarez F, Ortega R, Gomez-Polo C, Barmak AB, Kois JC, Revilla-Leon M. Influence of the implant scan body bevel location, implant angulation and position on intraoral scanning accuracy: An in vitro study. J Dent. 2022 Jun;121:104122. doi: 10.1016/j.jdent.2022.104122. Epub 2022 Apr 6. PMID 35395345
- [Background] Lin WS, Harris BT, Elathamna EN, Abdel-Azim T, Morton D. Effect of implant divergence on the accuracy of definitive casts created from traditional and digital implant-level impressions: an in vitro comparative study. Int J Oral Maxillofac Implants. 2015 Jan-Feb;30(1):102-9. doi: 10.11607/jomi.3592. PMID 25615919
- [Background] Carneiro Pereira AL, Medeiros VR, da Fonte Porto Carreiro A. Influence of implant position on the accuracy of intraoral scanning in fully edentulous arches: A systematic review. J Prosthet Dent. 2021 Dec;126(6):749-755. doi: 10.1016/j.prosdent.2020.09.008. Epub 2020 Oct 23. PMID 33268069
- [Background] Basaki K, Alkumru H, De Souza G, Finer Y. Accuracy of Digital vs Conventional Implant Impression Approach: A Three-Dimensional Comparative In Vitro Analysis. Int J Oral Maxillofac Implants. 2017 July/August;32(4):792-799. doi: 10.11607/jomi.5431. Epub 2017 Jun 14. PMID 28618432
- [Background] Revilla-Leon M, Kois DE, Kois JC. A guide for maximizing the accuracy of intraoral digital scans. Part 1: Operator factors. J Esthet Restor Dent. 2023 Jan;35(1):230-240. doi: 10.1111/jerd.12985. Epub 2022 Dec 7. PMID 36479807
- [Background] Revilla-Leon M, Kois DE, Kois JC. A guide for maximizing the accuracy of intraoral digital scans: Part 2-Patient factors. J Esthet Restor Dent. 2023 Jan;35(1):241-249. doi: 10.1111/jerd.12993. Epub 2023 Jan 13. PMID 36639916
- [Background] Revilla-Leon M, Gohil A, Barmak AB, Gomez-Polo M, Perez-Barquero JA, Att W, Kois JC. Influence of ambient temperature changes on intraoral scanning accuracy. J Prosthet Dent. 2023 Nov;130(5):755-760. doi: 10.1016/j.prosdent.2022.01.012. Epub 2022 Feb 21. PMID 35210107
- [Background] Revilla-Leon M, Subramanian SG, Ozcan M, Krishnamurthy VR. Clinical Study of the Influence of Ambient Light Scanning Conditions on the Accuracy (Trueness and Precision) of an Intraoral Scanner. J Prosthodont. 2020 Feb;29(2):107-113. doi: 10.1111/jopr.13135. Epub 2019 Dec 30. PMID 31860144
- [Background] Revilla-Leon M, Subramanian SG, Att W, Krishnamurthy VR. Analysis of Different Illuminance of the Room Lighting Condition on the Accuracy (Trueness and Precision) of An Intraoral Scanner. J Prosthodont. 2021 Feb;30(2):157-162. doi: 10.1111/jopr.13276. Epub 2020 Nov 7. PMID 33094878
- [Background] Revilla-Leon M, Jiang P, Sadeghpour M, Piedra-Cascon W, Zandinejad A, Ozcan M, Krishnamurthy VR. Intraoral digital scans: Part 2-influence of ambient scanning light conditions on the mesh quality of different intraoral scanners. J Prosthet Dent. 2020 Nov;124(5):575-580. doi: 10.1016/j.prosdent.2019.06.004. Epub 2019 Dec 20. PMID 31870612
- [Background] Revilla-Leon M, Jiang P, Sadeghpour M, Piedra-Cascon W, Zandinejad A, Ozcan M, Krishnamurthy VR. Intraoral digital scans-Part 1: Influence of ambient scanning light conditions on the accuracy (trueness and precision) of different intraoral scanners. J Prosthet Dent. 2020 Sep;124(3):372-378. doi: 10.1016/j.prosdent.2019.06.003. Epub 2019 Dec 19. PMID 31864638
- [Background] Abduo J, Lyons K, Bennani V, Waddell N, Swain M. Fit of screw-retained fixed implant frameworks fabricated by different methods: a systematic review. Int J Prosthodont. 2011 May-Jun;24(3):207-20. PMID 21519567
- [Background] Abduo J, Bennani V, Waddell N, Lyons K, Swain M. Assessing the fit of implant fixed prostheses: a critical review. Int J Oral Maxillofac Implants. 2010 May-Jun;25(3):506-15. PMID 20556249
- [Background] Katsoulis J, Takeichi T, Sol Gaviria A, Peter L, Katsoulis K. Misfit of implant prostheses and its impact on clinical outcomes. Definition, assessment and a systematic review of the literature. Eur J Oral Implantol. 2017;10 Suppl 1:121-138. PMID 28944373
- [Background] Jemt T. Failures and complications in 391 consecutively inserted fixed prostheses supported by Branemark implants in edentulous jaws: a study of treatment from the time of prosthesis placement to the first annual checkup. Int J Oral Maxillofac Implants. 1991 Fall;6(3):270-6. PMID 1813395
- [Background] Klineberg IJ, Murray GM. Design of superstructures for osseointegrated fixtures. Swed Dent J Suppl. 1985;28:63-9. No abstract available. PMID 3904064
- [Background] Mangano F, Gandolfi A, Luongo G, Logozzo S. Intraoral scanners in dentistry: a review of the current literature. BMC Oral Health. 2017 Dec 12;17(1):149. doi: 10.1186/s12903-017-0442-x. PMID 29233132
- [Background] Flugge TV, Att W, Metzger MC, Nelson K. Precision of Dental Implant Digitization Using Intraoral Scanners. Int J Prosthodont. 2016 May-Jun;29(3):277-83. doi: 10.11607/ijp.4417. PMID 27148990
- [Background] Wismeijer D, Joda T, Flugge T, Fokas G, Tahmaseb A, Bechelli D, Bohner L, Bornstein M, Burgoyne A, Caram S, Carmichael R, Chen CY, Coucke W, Derksen W, Donos N, El Kholy K, Evans C, Fehmer V, Fickl S, Fragola G, Gimenez Gonzales B, Gholami H, Hashim D, Hui Y, Kokat A, Vazouras K, Kuhl S, Lanis A, Leesungbok R, van der Meer J, Liu Z, Sato T, De Souza A, Scarfe WC, Tosta M, van Zyl P, Vach K, Vaughn V, Vucetic M, Wang P, Wen B, Wu V. Group 5 ITI Consensus Report: Digital technologies. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:436-442. doi: 10.1111/clr.13309. PMID 30328201
- [Background] Kim JH, Kim KR, Kim S. Critical appraisal of implant impression accuracies: A systematic review. J Prosthet Dent. 2015 Aug;114(2):185-92.e1. doi: 10.1016/j.prosdent.2015.02.005. Epub 2015 Apr 30. PMID 25935089
- [Background] Lee SJ, Gallucci GO. Digital vs. conventional implant impressions: efficiency outcomes. Clin Oral Implants Res. 2013 Jan;24(1):111-5. doi: 10.1111/j.1600-0501.2012.02430.x. Epub 2012 Feb 22. PMID 22353208
- [Background] Tabesh M, Nejatidanesh F, Savabi G, Davoudi A, Savabi O, Mirmohammadi H. Marginal adaptation of zirconia complete-coverage fixed dental restorations made from digital scans or conventional impressions: A systematic review and meta-analysis. J Prosthet Dent. 2021 Apr;125(4):603-610. doi: 10.1016/j.prosdent.2020.01.035. Epub 2020 Apr 10. PMID 32284188
- [Background] Revilla-Leon M, Frazier K, da Costa JB, Kumar P, Duong ML, Khajotia S, Urquhart O; Council on Scientific Affairs. Intraoral scanners: An American Dental Association Clinical Evaluators Panel survey. J Am Dent Assoc. 2021 Aug;152(8):669-670.e2. doi: 10.1016/j.adaj.2021.05.018. PMID 34325781
- [Background] Alghazzawi TF. Advancements in CAD/CAM technology: Options for practical implementation. J Prosthodont Res. 2016 Apr;60(2):72-84. doi: 10.1016/j.jpor.2016.01.003. Epub 2016 Feb 28. PMID 26935333
- [Background] Watanabe H, Fellows C, An H. Digital Technologies for Restorative Dentistry. Dent Clin North Am. 2022 Oct;66(4):567-590. doi: 10.1016/j.cden.2022.05.006. Epub 2022 Sep 11. PMID 36216447
- [Background] Wang J, Wang B, Liu YY, Luo YL, Wu YY, Xiang L, Yang XM, Qu YL, Tian TR, Man Y. Recent Advances in Digital Technology in Implant Dentistry. J Dent Res. 2024 Jul;103(8):787-799. doi: 10.1177/00220345241253794. Epub 2024 May 31. PMID 38822563